CLINICAL TRIAL: NCT05207007
Title: Visual Function in Pediatric Patients With Posterior Polar Cataracts and Posterior Lenticonus
Brief Title: Visual Function in Pediatric Patients With Posterior Lens Opacities
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Childhood Cataract Program of the Chinese Ministry of Health(CCPMOH), Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: CCPMOH2020-China20
Record Dates: First submitted 2022-01-09; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Congenital Cataract Polar Posterior
Keywords: visual function; posterior polar cataracts; posterior lenticonus
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- posterior polar cataracts: Phacomulsification lens removal cataract surgery with Intraocular lens(IOL) implantation were performed in these patients.
  Drug: Subconjunctival dexamethasone and general anesthesia All patients received subconjunctival dexamethasone (2 mg) during surgery, and all surgeries were performed under general anesthesia.
  Interventions: Procedure: Phacomulsification lens removal cataract surgery with Intraocular lens(IOL) implantation
- posterior lenticonus: Phacomulsification lens removal cataract surgery with Intraocular lens(IOL) implantation were performed in these patients.
  Drug: Subconjunctival dexamethasone and general anesthesia All patients received subconjunctival dexamethasone (2 mg) during surgery, and all surgeries were performed under general anesthesia.
  Interventions: Procedure: Phacomulsification lens removal cataract surgery with Intraocular lens(IOL) implantation

INTERVENTIONS:
Procedure: Phacomulsification lens removal cataract surgery with Intraocular lens(IOL) implantation — Phacomulsification lens removal cataract surgery with IOL implantation in both two groups

SUMMARY:
Prognostic factors determining visual outcomes in patients with posterior polar cataracts and posterior lenticonus are largely unknown. In this trial, the investigators aimed to evaluate the visual outcomes in patients with posterior polar cataracts and posterior lenticonus and try to find out the factors associated with the visual acuity after surgery. Patients enrolled in this study will be followed for at least 6 months and will have study visits at 1 day, 1 week, 1 month, 3 month, 6 month postoperatively.

DETAILED DESCRIPTION:
Congenital cataract patients have a wide range of presentations of lens opacities with different impact on visual function. Polar cataracts are opacities of the subcapsular cortex in the polar regions of the lens. To our knowledge, anterior polar cataracts are usually visually insignificant, however, even a small posterior lens opacity can impair vision because of their close proximity to the macula. Visual impairment could be caused by an opacity that blocks the visual axis, refractive error, posterior lesion-induced optical distortion, or amblyopia. Therefore, surgery is often recommended when visual function is significantly affected. The primary indication for surgical intervention in cataract is poor visual acuity. However, the previous studies have shown that preoperative visual acuity is a poor predictor of improvement in the subjectively experienced quality of vision after cataract surgery. Considering the increased risk for capsule rupture during surgery and the sacrifice of accommodation after cataract surgery in eyes with posterior lens opacities, the decision of surgical intervention must be carefully weighed.

In this trial, the investigators aimed to evaluate the changes of visual function, including visual acuity, modulation transfer function, ocular aberrations in the participants with posterior lens opacities. Moreover, various factors which might be associated with postoperative visual acuity were explored. The participants enrolled in this study will be followed for at least 6 months and will have study visits at 1 day, 1 week, 1 month, 3 month, 6 month postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Children with posterior polar cataracts or posterior lenticonus who need cataract surgery
* Aged 3-14 years
* Have signed a consent form
* Can be followed

Exclusion Criteria:

* Have relevant ocular disease other than congenital cataract
* Could not cooperate to the examinations

Ages: 3 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Patients with congenital posterior polar cataracts or posterior lenticonus who need cataract surgery at the Zhongshan Ophthalmic Center, Sun Yat-sen University in China were included. The patients who had relevant ocular disease other than congenital cataract or could not cooperate to the examinations were excluded. The indication for surgery in all patients was significantly deteriorated visual function and amblyopia treatment failure (decline in CDVA to 20/80 or worse). The study adhered to the tenets of the Declaration of Helsinki. Written informed consent was obtained from each subject.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-01-04 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
Visual acuity (BCVA) | 6 month after surgery
  Visual acuity (BCVA) measured by ETDRS chart after surgery
Stereoacuity | 6 month after surgery
  Stereoacuity measured at 40 cm using the Randot stereotests
modulation transfer function (MTF) | 6 month after surgery
  MTF measured with the Optical Quality Analysis System
monochromatic aberrations | 6 month after surgery
  monochromatic aberrations measured by the iTrace Dynamic Laser Refraction

SECONDARY OUTCOMES:
Location of the cataracts | before surgery
  divided into central, paracentral, and peripheral
size of lens lesion | before surgery
  measured by image J
Visual acuity (BCVA) | before surgery
  Visual acuity (BCVA) measured by ETDRS chart before surgery
Stereoacuity | before surgery
  Stereoacuity measured at 40 cm using the Randot stereotests
modulation transfer function (MTF) | before surgery
  MTF measured with the Optical Quality Analysis System
monochromatic aberrations | before surgery
  monochromatic aberrations measured by the iTrace Dynamic Laser Refraction system

CONTACTS AND LOCATIONS:
Overall Officials: Weirong Chen, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No